CLINICAL TRIAL: NCT00424099
Title: A Randomized Controlled Trial of Methylphenidate and a Nursing Telephone Intervention (NTI) for Fatigue in Advanced Cancer Patients
Brief Title: Methylphenidate and a Nursing Telephone Intervention for Fatigue
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2005-0613; R01NR010162-01A1 (NIH); NCI-2012-01571 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Advanced Cancer; Fatigue
Keywords: Advanced Cancer; Fatigue; Nursing Telephone Intervention; NTI; Methylphenidate; Placebo; Ritalin
MeSH Terms: conditions — Fatigue | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Methylphenidate + NTI (Experimental): Methylphenidate 5 mg (one capsule) orally every two hours as needed up to a maximum of 20 mg per day for a period of 14 days + Nursing Telephone Intervention (NTI). NTI calls from study nurse 3 times weekly to ask about side effects and other symptoms.
  Interventions: Drug: Methylphenidate; Behavioral: Nursing Telephone Intervention
- Group 2: Placebo + NTI (Placebo Comparator): Placebo capsule orally as needed for 14 days + NTI, calls from study nurse 3 times weekly to ask about side effects and other symptoms.
  Interventions: Behavioral: Nursing Telephone Intervention; Drug: Placebo
- Group 3: Methylphenidate + Non NTI (Experimental): Methylphenidate 5 mg (one capsule) orally every two hours as needed up to a maximum of 20 mg per day for a period of 14 days + Non NTI, calls from research staff 3 times weekly.
  Interventions: Drug: Methylphenidate; Behavioral: Non NTI
- Group 4: Placebo + Non NTI (Experimental): Placebo capsules as needed with Non NTI, calls from research staff 3 times weekly.
  Interventions: Drug: Placebo; Behavioral: Non NTI

INTERVENTIONS:
Drug: Methylphenidate — 5 mg (one capsule) orally every two hours as needed up to a maximum of 20 mg per day for a period of 14 days.
  Other Names: Ritalin
  Arms: Group 1: Methylphenidate + NTI; Group 3: Methylphenidate + Non NTI
Behavioral: Nursing Telephone Intervention — Call from study nurse 3 times weekly to ask about side effects and other symptoms.
  Other Names: NTI
  Arms: Group 1: Methylphenidate + NTI; Group 2: Placebo + NTI
Drug: Placebo — One capsule, orally every two hours as needed up to a maximum of 4 capsules per day for a period of 14 days.
  Arms: Group 2: Placebo + NTI; Group 4: Placebo + Non NTI
Behavioral: Non NTI — Non NTI are calls from research staff 3 times weekly.
  Other Names: Non Nursing Telephone Intervention
  Arms: Group 3: Methylphenidate + Non NTI; Group 4: Placebo + Non NTI

SUMMARY:
The goal of this clinical research study is to learn if methylphenidate (Ritalin) can help to control fatigue caused by cancer. Its effect on other symptoms such as drowsiness, depression, sleeplessness, physical activity, and anxiety will also be studied. Another goal of this study is to learn if receiving a phone call by a nurse improves fatigue in patients.

DETAILED DESCRIPTION:
Fatigue is one of the most common problems in patients with advanced cancer. Currently, there are no treatments for managing fatigue. Methylphenidate is a stimulant that increases ability to pay attention, increases mental alertness, and decreases feelings of fatigue.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to one of 4 groups. You will have an equal chance of being placed in any of the 4 groups. You, the medical staff, and researchers will not know to which group you have been assigned.

Regardless of which group you are in, you will record your fatigue in a daily diary at breakfast, lunch, dinner, and before bedtime. Based on your level of fatigue, you will take the study drug as needed. You can take the study drug every 2 hours but you may not take more than 4 capsules a day.

Participants in Group 1 will take a methylphenidate capsule by mouth as needed to relieve symptoms of fatigue for 14 days. A nurse will call you 4-6 times in the first two weeks to ask about side effects and other symptoms. The phone calls should take about 10-20 minutes. The study nurse will set up a convenient time for you to take the phone call.

Participants in Group 2 will take a placebo capsule by mouth as needed for 14 days. A placebo is a capsule that does not contain any medication but looks just like the methylphenidate. A nurse will call you 4-6 times in the first two weeks to ask about side effects and other symptoms. The phone calls should take about 10-20 minutes. The study nurse will set up a convenient time for you to take the phone call.

Participants in Group 3 will take a methylphenidate capsule by mouth as needed for 14 days. Participants in this group will not receive any calls from a study nurse. However, A research staff member will call you 4-6 times in the first two weeks to ask about side effects and other symptoms. The phone calls should take about 10-20 minutes. The research staff member will set up a convenient time for you to take the phone call.

Participants in Group 4 will take a placebo capsule by mouth as needed for 14 days. Participants in this group will not receive any calls from a study nurse. However, A research staff member will call you 4-6 times in the first two weeks to ask about side effects and other symptoms. The phone calls should take about 10-20 minutes. The research staff member will set up a convenient time for you to take the phone call.

You will be asked to wear a wrist actigraph monitor (a wristwatch that keeps track of your physical activity and your sleep cycles) for the first 14 days.

You will keep a daily diary of your fatigue and other symptoms, the number and times pills are taken, and your fatigue rating before and 2 hours after taking methylphenidate.

On about day 15 (or within 3 days) you will return to the palliative care clinic at M. D. Anderson for tests. You will be asked about your level of drowsiness, pain, constipation, and fatigue. You will be asked about any side effects you may have experienced and the effectiveness of the drug. You will repeat the 6 minute physical test, the cognitive status test, and you will return the actigraph monitor to the research nurse. You will also be given the option to receive up to 4 capsules of methylphenidate per day until Day 36. You will not be told whether you were taking placebo or methylphenidate during Days 1-14. If you cannot come to the clinic on Day 15, all tests except the walking test, may be performed over the telephone. You will be asked to mail the actigraph back.

If you decide not to take methylphenidate on Days 15-36, you will be considered off-study and you will have end-of-study tests on Day 15. If you decide to take methylphenidate on Days 15-36, you will remain on study until Day 36. On Day 36, you will have end-of-study tests.

For end-of-study tests, you will repeat the physical and cognitive tests. You will be asked about your symptoms and any side effects you may be experiencing. You will then return to your primary physician who will discuss with you whether or not to continue on the methylphenidate based on your response to the drug.

Your participation in this study should end on either Day 15 or Day 36. However, if you develop intolerable side effects (including fatigue) while on this study, the medication will be stopped and you will be removed from the study.

This is an investigational study. Methylphenidate has been approved by the FDA and is a commercially available drug. It is FDA approved at this dose level. Its use in this study, for this purpose, is investigational. About 212 patients will take part in this multicenter study. About 142 patients will be enrolled at The University of Texas (UT) MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be eligible to participate in this study if they have advanced cancer.
2. Patients will be eligible to participate in this study if they rate fatigue on the Edmonton Symptom Assessment System (ESAS) during the last 24 hours as greater than or equal to 4 on a 0-10 scale, in which 0= no fatigue and 10=worst possible fatigue
3. Describe fatigue as being present every day for most of day for a minimum of 2 weeks
4. Lack clinical evidence of cognitive failure, with normal Mini Mental State Examination (MMSE). A score of 24 is considered normal
5. Are 18 years or older
6. Are willing to keep a daily diary, engage in telephone follow up with a nurse every other day, and return for follow-up visit after 14 days of treatment
7. Have telephone access to be contacted by the research nurse. If patient is relocating within 5 weeks, patient will be asked to provide a new telephone number
8. Hemoglobin of greater than or equal to 8 g/dl within 2 weeks of enrollment. If the patient has not had blood drawn for a hemoglobin level in the past 2 weeks, one will be done to determine the eligibility. Patients with a hemoglobin of less than 8 will be referred for treatment of their anemia
9. Able to understand the description of the study and give written informed consent.
10. Able to understand the description of assessments, and able to complete baseline assessment
11. Patients on no erythropoietin or stable dose.

Exclusion Criteria:

1. Major contraindication to methylphenidate i.e. hypersensitivity, anxiety, tension, agitation, or motor tics, glaucoma, severe angina pectoris, or hypertension, etc.
2. Currently on methylphenidate or has been on methylphenidate within the last 10 days.
3. Inability to complete the baseline assessment forms or do understand the recommendations for participation in the study
4. Major depression according to the Structured Clinical Interview (SCID) Diagnostic and Statistical Manual of Mental Disorders (DSM) IV diagnostic criteria. These patients wil be referred immediately to psychiatry for assessment and management
5. Pregnant or lactating women
6. Requirement for Monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants or clonidine
7. Glaucoma, history of marked anxiety disorders
8. History of alcohol (CAGE questionnaire score for the last 2 years is 2 or above on a 0 to 4 scale) or substance abuse including illegal drugs and/or medications.
9. Tourette's syndrome
10. Symptomatic tachycardia and uncontrolled hypertension.
11. Currently receiving oral anticoagulants (Coumadin/warfarin), anticonvulsants (Phenobarbital, diphenylhydantoin, primidone), phenylbutazone, and tricyclic drugs (imipramine, clomipramine, desipramine).
12. Patients with pacemakers
13. Patients with symptomatic cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2007-01-09 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson (LBJ) Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Yennurajalingam S, Tayjasanant S, Balachandran D, Padhye NS, Williams JL, Liu DD, Frisbee-Hume S, Bruera E. Association between Daytime Activity, Fatigue, Sleep, Anxiety, Depression, and Symptom Burden in Advanced Cancer Patients: A Preliminary Report. J Palliat Med. 2016 Aug;19(8):849-56. doi: 10.1089/jpm.2015.0276. Epub 2016 May 5. PMID 27148765
- [Derived] Bruera E, Yennurajalingam S, Palmer JL, Perez-Cruz PE, Frisbee-Hume S, Allo JA, Williams JL, Cohen MZ. Methylphenidate and/or a nursing telephone intervention for fatigue in patients with advanced cancer: a randomized, placebo-controlled, phase II trial. J Clin Oncol. 2013 Jul 1;31(19):2421-7. doi: 10.1200/JCO.2012.45.3696. Epub 2013 May 20. PMID 23690414
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from outpatient palliative care and oncology clinics at MD Anderson Cancer Center or from outpatient clinics at Lyndon B. Johnson General Hospital in Houston, Texas.
Pre-assignment Details: A total of 197 participants were enrolled in the study but 190 were randomized. 7 participants were not randomized for various reasons.
Groups:
- Methylphenidate (MP) + Nursing Telephone Intervention (NTI): One 5-mg Methylphenidate capsule was administered orally every 2 hours as needed up to 20 mg per day for 14 days and NTI phone calls four to six times over the 2 weeks
- Methylphenidate (MP) + Control Telephone Intervention (CTI): One 5-mg Methylphenidate capsule was administered orally every 2 hours as needed up to 20 mg per day for 14 days and CTI phone calls four to six times over the 2 weeks
- Placebo (PL)+ Nursing Telephone Intervention (NTI): One Placebo capsule was administered orally every 2 hours as needed up to four capsules per day for 14 days and NTI phone calls four to six times over the 2 weeks
- Placebo (PL) + Control Telephone Intervention (CTI): One Placebo capsule was administered orally every 2 hours as needed up to four capsules per day for 14 days and CTI phone calls four to six times over the 2 weeks
Period: Overall Study
Arm/Group | Methylphenidate (MP) + Nursing Telephone Intervention (NTI) | Methylphenidate (MP) + Control Telephone Intervention (CTI) | Placebo (PL)+ Nursing Telephone Intervention (NTI) | Placebo (PL) + Control Telephone Intervention (CTI)
Started | 45 | 47 | 50 | 48
Completed | 38 | 31 | 38 | 35
Not Completed | 7 | 16 | 12 | 13
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Illness | 2 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0
Not completed — Hospitalized | 1 | 2 | 1 | 3
Not completed — UNABLE OR Unavailable to complete questionnaires | 3 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 9 | 4 | 6
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Missing | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analyses included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate (MP) + Nursing Telephone Intervention (NTI) | Methylphenidate (MP) + Control Telephone Intervention (CTI) | Placebo (PL)+ Nursing Telephone Intervention (NTI) | Placebo (PL) + Control Telephone Intervention (CTI) | Total
Number analyzed (Participants) | 45 | 47 | 50 | 48 | 190
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 83] | 56 [32 to 84] | 59 [32 to 84] | 58 [52 to 83] | 57.5 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 33 | 32 | 128
  Male | 16 | 13 | 17 | 16 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 10 | 8 | 32
  Not Hispanic or Latino | 37 | 41 | 40 | 40 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 4 | 7 | 19
  White | 42 | 40 | 46 | 41 | 169
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 47 | 50 | 48 | 190
Baseline Functional Assessment of Chronic Illness Therapy (FACIT-F ) Fatigue Subscale Score [Median (Inter-Quartile Range); unit: score on a scale] — FACIT Fatigue Subscale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is from 0-52. The higher the score, the lower the fatigue level.
  score on a scale | 21.50 [15.00 to 27.00] | 20.00 [15.00 to 29.00] | 20.00 [12.00 to 25.00] | 21.50 [13.25 to 27.75] | 20.00 [14.00 to 27.00]
Baseline Edmonton Symptom Assessment System (ESAS) Fatigue Score [Median (Inter-Quartile Range); unit: score on a scale] — The Edmonton Symptom Assessment Scale (ESAS) is used to rate the intensity of ten common symptoms including fatigue experienced by cancer patients. The ESAS allows patients to rate the intensity of their fatigue using a 0-10 scale (0 = not at all, 10 = worst possible). The total ESAS score range from 0-100. The lower the score, the lower the fatigue level.
  score on a scale | 7.00 [5.00 to 8.00] | 6.00 [5.00 to 7.25] | 6.00 [5.00 to 7.25] | 6.00 [5.00 to 7.00] | 6.00 [5.00 to 8.00]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Fatigue Subscale Score
Description: FACIT-F fatigue subscale consists of 13 items. Patients rate the intensity of their fatigue symptoms on a scale of 0 to 4 (0=not at all and 4=very much). Total FACIT-F fatigue subscale score ranges from 0 to 52 with higher scores indicate higher fatigue. We measured the median change in FACIT-F fatigue sub scale score between Baseline and Day 15 using Kruskal-Wallis test.
Time Frame: Baseline and Day 15
Population: Those who completed intervention up to day 15
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methylphenidate (MP) + Nursing Telephone Intervention (NTI) | Methylphenidate (MP) + Control Telephone Intervention (CTI) | Placebo (PL)+ Nursing Telephone Intervention (NTI) | Placebo (PL) + Control Telephone Intervention (CTI)
Number analyzed (Participants) | 37 | 31 | 38 | 35
score on a scale | 4.00 [-2.00 to 11.0] | 7.00 [2.00 to 11.00] | 8.50 [3.00 to 17.00] | 5.00 [0.00 to 6.00]
Statistical Analysis 1: Comparison: Methylphenidate (MP) + Nursing Telephone Intervention (NTI) vs Methylphenidate (MP) + Control Telephone Intervention (CTI) vs Placebo (PL)+ Nursing Telephone Intervention (NTI) vs Placebo (PL) + Control Telephone Intervention (CTI); Test type: Other; p = 0.16, Kruskal-Wallis

2. Secondary Outcome: Change in Edmonton Symptom Assessment System (ESAS) Fatigue Score
Description: The ESAS was used to assess the following 9 symptoms commonly experienced symptoms by cancer patients: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, and well-being. Patients rate the intensity of their fatigue symptoms on a scale of 0 to 10 (0=not at all and 10=very much). Total ESAS fatigue score ranges from 0 to 10 with higher scores indicate higher fatigue. We measured the median change in ESAS fatigue score between Baseline and Day 15 using Kruskal-Wallis test.
Time Frame: Baseline and Day 15
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methylphenidate (MP) + Nursing Telephone Intervention (NTI) | Methylphenidate (MP) + Control Telephone Intervention (CTI) | Placebo (PL)+ Nursing Telephone Intervention (NTI) | Placebo (PL) + Control Telephone Intervention (CTI)
Number analyzed (Participants) | 37 | 29 | 37 | 34
score on a scale | -3.00 [-4.00 to -1.00] | -1.00 [-3.00 to 0] | -2.00 [-5.00 to 0] | -2.00 [-4.00 to 0]
Statistical Analysis 1: Comparison: Methylphenidate (MP) + Nursing Telephone Intervention (NTI) vs Methylphenidate (MP) + Control Telephone Intervention (CTI) vs Placebo (PL)+ Nursing Telephone Intervention (NTI) vs Placebo (PL) + Control Telephone Intervention (CTI); Test type: Other; p = 0.45, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse events measured up to 15 days
Description: Adverse Events data were presented in 2 arms. The reason is that only the Intervention medicine Methylphenidate (MP) can produce Adverse Events, not the telephone calls.
  This is why the two Methylphenidate arms (MP+ NTI and MP+CTI) were combined into one arm and similarly the two Placebo arms were combined into one arm.
Groups:
- Methylphenidate (MP) +Nursing Telephone Intervention (NTI): One 5-mg Methylphenidate capsule was administered orally every 2 hours as needed up to 20 mg per day for 14 days and NTI phone calls four to six times over the 2 weeks
- Methylphenidate (MP) +Control Telephone Intervention (CTI): One 5-mg Methylphenidate capsule was administered orally every 2 hours as needed up to 20 mg per day for 14 days and CTI phone calls four to six times over the 2 weeks
Arm/Group | Methylphenidate (MP) +Nursing Telephone Intervention (NTI) | Methylphenidate (MP) +Control Telephone Intervention (CTI) | Placebo (PL)+ Nursing Telephone Intervention (NTI) | Placebo (PL) + Control Telephone Intervention (CTI)
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/47 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 9/45 | 4/47 | 4/50 | 9/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (MP) +Nursing Telephone Intervention (NTI) (N=45) | Methylphenidate (MP) +Control Telephone Intervention (CTI) (N=47) | Placebo (PL)+ Nursing Telephone Intervention (NTI) (N=50) | Placebo (PL) + Control Telephone Intervention (CTI) (N=48)
Pain (Nervous system disorders) | 2 | 1 | 2 | 1
Insomnia (Nervous system disorders) | 3 | 0 | 1 | 3
Mood Alteration (Psychiatric disorders) | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1 | 0 | 1
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Syncope (Cardiac disorders) | 0 | 0 | 1 | 0
Flu-like symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Slurred Speech (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-02-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT00424099/Prot_SAP_000.pdf